CLINICAL TRIAL: NCT03807830
Title: Exploring the Use of ECochG Testing During Electrode Insertion in Cochlear Implant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Sophie Newton, Hearing implant nurse. Prof M Bance Chief Investigator., Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18/EE/0304
Record Dates: First submitted 2019-01-11; First posted 2019-01-17 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Cochlear Implants; Hearing Preservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm feasbility study (Other)
  Interventions: Procedure: Electrocochlography

INTERVENTIONS:
Procedure: Electrocochlography — Intra-operative ECochG recording via the implant, post operative ECochG measurements. Impedances measured over time.

SUMMARY:
Investigation of a new ECoChG system (Electrocochleography) during the surgical insertion of cochlear implants, for patients with Advanced Bionics devices.

The sound recordings created may be useful in aiding the surgeon to better implant the patient by letting him or her know if they are damaging the ear during implantation in real time

Patients will be followed up for 1 year post surgery within our trial, and have a further 3 ECochGs performed in the clinic setting, (6 weeks, 6 months, 1 year) through their implants.

DETAILED DESCRIPTION:
Cochlear implant candidature has changed in the past years. Today many cochlear implant recipients have some low frequency residual hearing in the ear which is to be implanted. To help preserve hearing, the electrode array must be inserted extremely carefully. It is desirable to have real-time feedback relating to progress of the electrode insertion.

One possible tool that might provide this is an electrocochleography (ECochG). A brief low-frequency acoustic tone at a fixed level is delivered to the external ear canal. This results in normal movements of the outer and the inner hair cells inside the inner ear. These movements are known to produce small electrical potentials that have been previously been sensed by a recording electrode placed on the promontory, or surface of the bone in which the cochlea is located. Averaging of these recordings in synchrony with the acoustic stimulus allows the small ECochG signal to be reinforced while any physiological or electrical noise is averaged out. With ECochG measurements different aspects of the auditory system can be tested. For the investigators work only the cochlear microphonic, generated by the outer hair cells will be recorded and analysed.

The Advanced Bionics (AB) implant system is uniquely suited to do such measurements. The aim of the study is to monitor electrode array insertion during surgery and any residual hearing function over time in using this tool as a comparison to conventional methods. Subjects will undergo the study procedure of ECochG measurements, alongside additional standard of care appointments for the research, pure tone audiometry and impedence measurement. Only a 10 minute ECochG measurement will be the additional research component to the patients clinical routine as mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Patients between ages of 12 months to 6 years old, and Adults over 18 years old
* Meets normal candidacy requirements for cochlear implantation
* Advanced Bionics (AB) implant has been selected for patient at MDT
* Patient has capacity to consent
* Patent cochlea as verified by CT or MRI scan
* No cochlear abnormality that might prevent insertion of the electrode array
* Measurable residual hearing in the ear to be implanted
* No additional handicap that would prevent study procedures being followed
* Agreement to participate in the study

Exclusion Criteria:

* Complex cases where minimal duration of surgery is required. Although ECochG adds less than 10 minutes to the surgery time.
* Patients lacking the capacity to consent

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Measure cochlear micro phonic amplitude | 12 months
  To measure objectively the cochlear micro phonic amplitude either intra or post operatively within initial 12 months of cochlear implant use

CONTACTS AND LOCATIONS:
Overall Officials: Manohar L Bance, MD, Principal Investigator — The Emmeline Centre for Cochlear Implants
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided